CLINICAL TRIAL: NCT05191823
Title: Long-term Effects and Safety of DHA+AA Supplementation in Toddlerhood for Children Born Preterm
Brief Title: Omega Tots Long Term Follow-up
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Keim (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Sarah Keim, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00001037; R01HD100493 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Preterm Birth; Child Development
MeSH Terms: conditions — Premature Birth | interventions — Docosahexaenoic Acids; Arachidonic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docosahexaenoic Acid + Arachidonic Acid (Experimental): Docosahexaenoic Acid + Arachidonic Acid (DHA+AA)
  Interventions: Drug: Docosahexaenoic Acid + Arachidonic Acid (DHA+AA)
- Placebo (Placebo Comparator): Corn oil supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Docosahexaenoic Acid + Arachidonic Acid (DHA+AA) — 200 mg DHA+ 200 mg AA per day for 6 months
  Arms: Docosahexaenoic Acid + Arachidonic Acid
Dietary Supplement: Placebo — 400 mg corn oil per day for 6 months
  Arms: Placebo

SUMMARY:
This is a continuation study to the Omega Tots trial (NCT01576783). The purpose of this study is to follow-up with participants of the original study to determine the long-term effect a daily fatty acid dietary supplement taken during toddlerhood might have on children born preterm now that they are 8.5-10.5 years old.

DETAILED DESCRIPTION:
The overall objective with the present study is to determine the long-term effects of docosahexaenoic acid (DHA) plus arachidonic acid (AA) supplementation on general cognitive ability, language, and executive function, and to examine genetic explanations for treatment effects, through one comprehensive study visit with children and parents from the Omega Tots trial cohort (NCT01576783).

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in Omega Tots (NCT01576783).
* Current age of 8 years, 180 days to 10 years, 180 days.

Exclusion Criteria:

* Child in custody of children's services for their window of eligibility

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
General Cognitive Ability Score(Differential Ability Scales, Second Edition-DAS-II) | A single study visit when the child is between 8.5 years to 10.5 years
  Differential Ability Scales-II General Conceptual Ability assessment is a measure of general cognitive ability and is used to assess and identify children's cognitive strengths and weaknesses. The general cognitive ability score has a range from 30 to 170 (mean=100; SD=15). A low score indicates poor performance, and a high score indicates best performance.
Core Language Score (Clinical Evaluation of Language Fundamentals, Fifth edition-CELF-5) | A single study visit when the child is between 8.5 years to 10.5 years
  Clinical evaluation of Language Fundamentals, 5th edition core tests is a comprehensive measure of language and can assess children's written and oral language skills, as well as their reading comprehension. The core language score has a range from 30 to 170 (mean=100; SD=15). A low score indicates poor performance, and a high score indicates best performance.
Executive Function (NIH Toolbox) | A single study visit when the child is between 8.5 years to 10.5 years
  The NIH Toolbox Cognition Battery is a multi-dimensional set of brief measures assessing cognitive function. The Flanker, Dimensional Card Sort, and Pattern Comparison subtests measure executive function, processing speed, and attention. Standard scores have a range from 30 to 170 (mean=100; SD=15). A low score indicates poor performance, and a high score indicates best performance..

SECONDARY OUTCOMES:
Grooved Pegboard Task | A single study visit when the child is between 8.5 years to 10.5 years
  The Grooved Pegboard task measures eye-hand coordination and motor speed by requiring children to insert pegs into a board. The score is the time to place the pegs. If the child reaches the time limit of 3 minutes, then the score is the number of pegs placed. A faster time and lower number of pegs dropped is indicative of better performance.
Select subtest from the Wechsler Intelligence Scales for Children, Fifth Edition (WISC-V) | A single study visit when the child is between 8.5 years to 10.5 years
  The Weschler Intelligence Scales for Children-V Digit Span and Picture Span subtests assess working memory. The working memory index composite score has a range from 30-170 (mean=100; SD=15). A low score indicates poor performance, and a high score indicates best performance.
Select subtests from the Kaufman Test of Educational Achievement, Third Edition (KTEA-3) | A single study visit when the child is between 8.5 years to 10.5 years
  The Kaufman Test of Educational Achievement-3 is an assessment of key academic skills. The Letter and Word Recognition, Math Computation, Object Naming Facility, and Associative Fluency Subtests measure children's reading, math, and written language skills. The standard score has a range from 30-170 (mean=100; SD=15). A low score indicates poor performance, and a high score indicates best performance.
Anthropometrics-Body Composition (height) | A single study visit when the child is between 8.5 years to 10.5 years
  To assess children's body composition, height (in centimeters) is measured. This is converted to a z score for age and sex based on Child Growth Standards from the World Health Organization. The z score indicates the number of standard deviations away from the mean. A z score of 0 is equal to the mean of a reference population (children the same age and sex). Values less than 0 indicate values lower than the reference population, while values greater than 0 indicate values higher than the reference population.
Anthropometrics-Body Composition (weight) | A single study visit when the child is between 8.5 years to 10.5 years
  To assess children's body composition, weight (in kilograms) is measured. This is converted to a z score for age and sex based on Child Growth Standards from the World Health Organization. The z score indicates the number of standard deviations away from the mean. A z score of 0 is equal to the mean of a reference population (children the same age and sex). Values less than 0 indicate values lower than the reference population, while values greater than 0 indicate values higher than the reference population.
Anthropometrics-Adiposity | A single study visit when the child is between 8.5 years to 10.5 years
  To assess children's adiposity, a bioelectric impedance is used to measure body fat percent. Child's height and weight will be combined to report BMI (kg/m^2). These measurements are converted to a z score for age and sex based on Child Growth Standards from the World Health Organization. The z score indicates the number of standard deviations away from the mean. A z score of 0 is equal to the mean of a reference population (children the same age and sex). Values less than 0 indicate values lower than the reference population, while values greater than 0 indicate values higher than the reference population.
Behavior Rating Inventory of Executive Function, 2nd edition (BRIEF-2) | A single study visit when the child is between 8.5 years to 10.5 years
  The Behavior Rating Inventory of Executive Function, 2nd ed., is completed by the child's caregiver and teacher to measure a range of executive functioning capabilities in children. The BRIEF-2 yields nine clinical scales that measure various aspects of executive function plus three broad indices: behavioral regulation, emotion regulation, and cognitive regulation. Scores are summed to obtain a Global Executive Composite Score that will be expressed as a t score (range= [35-90]; (mean=50; SD=10), where a higher score indicates greater dysregulation .
Select subscales from the Teacher Report Form 6-18 | A single study visit when the child is between 8.5 years to 10.5 years
  The Teacher Report Form (syndrome and DSM-Oriented subscales) is completed by the child's teacher to reflect on the child's behavior in the previous six months. Scores are summed to provide a total problems score. Scores are also computed to measure the following subscales: internalizing problems, externalizing problems, anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, aggression behavior, affective problems, anxiety problems, somatic problems, attention deficit/hyperactivity problems, oppositional defiant problems, conduct problems. Scores will be expressed as a t-score (range= [33-100]; mean=50; SD=10), where a lower score indicates a more optimal outcome.
Child Behavior Checklist 6-18 (CBCL) | A single study visit when the child is between 8.5 years to 10.5 years
  The Child Behavior Checklist is completed by the child' caregiver to reflect their child's behavior in the previous six months. Scores were summed to provide total competence and problem scores. Total competence scores will be expressed as a t-score (range= [20-100]; mean=50; SD=10), where a higher score reflects a more optimal outcome. Problem scores will be expressed as a t-score (range= [25,100]; mean=50; SD=10), where a lower score reflects a more optimal outcome.
National Survey of Children's Health Module | A single study visit when the child is between 8.5 years to 10.5 years
  The National Survey of Children's Health module captures child developmental and behavioral diagnoses and other major diagnoses via parent report . A binary variable will be formed to indicate if a child has been diagnosed with each condition.
Emotion Regulation Checklist | A single study visit when the child is between 8.5 years to 10.5 years
  The Emotion Regulation Checklist is completed by the child's caregiver to measure child's ability to manage their emotions. Scores are grouped and summed to yield two scales: Emotion Regulation (range=10-40) and Lability/Negativity (range=14-56). Higher scores on the Emotion Regulation scale indicates more ability to regulate, whereas higher scores on the Lability/Negativity scale reflect greater dysregulation .
NIH Toolbox Friendship Fixed Form | A single study visit when the child is between 8.5 years to 10.5 years
  The NIH Toolbox Friendship (Ages 8-17) Fixed Form is a 5-item questionnaire that measures peer relationships and assesses the quality of relationships with friends and other acquaintances over the past month. Scores will be expressed as a t-score (range= [16-68]; mean=50; SD=10), where a higher score indicates stronger peer relationships.
NIH Toolbox Positive Peer Interaction Parent Report Fixed Form | A single study visit when the child is between 8.5 years to 10.5 years
  The NIH Toolbox Positive Peer Interaction Form (Ages 3-12) is a 4-item questionnaire that measures child peer relationships via parent report. Scores will be expressed as a t-score (range= [-8-63] ; mean=50; SD=10), where a higher score indicates stronger peer relationships.
Child Sleep Habits Questionnaire-abbreviated measure | A single study visit when the child is between 8.5 years to 10.5 years
  The Child Sleep Habits Questionnaire-abbreviated measures child sleep pattern and behaviors via parent report. Parents are asked to report on the child's bedtime behavior, sleep duration, and behavior during sleep. Scores are summed to give the total sleep disturbance score (range 33-99). Scores are also grouped and summed to yield eight subscales that measure different aspects of sleep. A higher score is indicative of more sleep problems .

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Keim, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05191823/Prot_SAP_000.pdf